CLINICAL TRIAL: NCT04401423
Title: Randomized Controlled Trial of Angiotensin 1-7 (TXA127) for the Treatment of Severe COVID-19
Brief Title: TXA127 for the Treatment of Severe COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Constant Therapeutics LLC (Industry)
Responsible Party: Principal Investigator, Jeanine D'Armiento, Associate Professor of Medicine (in Anesthesiology), Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAT0535
Record Dates: First submitted 2020-05-21; First posted 2020-05-26 (Actual); Results first posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: COVID-19
Keywords: COVID-19; multi-organ failure; acute kidney injury
MeSH Terms: conditions — COVID-19; Multiple Organ Failure; Acute Kidney Injury | interventions — angiotensin I (1-7)

STUDY DESIGN:
Intervention Model Description: Double-blinded, placebo-control, randomized clinical trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- TXA127 (Experimental): Participants will receive one 3-hour dosage (0.5 mg/kg per day), intravenously, for 10 days consecutively (or until discharge if less than 10 days).
  Interventions: Drug: TXA127
- Placebo (Placebo Comparator): Participants will receive one 3-hour dosage (0.5 mg/kg per day), intravenously, for 10 days consecutively (or until discharge if less than 10 days).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TXA127 — 0.5 mg/kg per day
  Other Names: angiotensin-(1-7)
  Arms: TXA127
Drug: Placebo — 0.5 mg/kg per day
  Other Names: control
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if administration of angiotensin-(1-7) (TXA127) prevents acute kidney injury and deterioration into multi-organ failure in patients with severe COVID-19. Participants will undergo a 10-day treatment with either placebo or study drug. The drug will be administered intravenously for 3 hours once each day for 10 days consecutively.

DETAILED DESCRIPTION:
Corona virus disease 2019 (COVID-19) has been associated with severe respiratory and multiorgan failure. Research shows that COVID-19 reduces levels of angiotensin-converting enzyme-2 (ACE-2), an enzyme that converts angiotensin II to angiotensin 1-7 (known as TXA127). COVID-19 reduces levels of ACE-2 and therefore angiotensin 1-7 and as a result, angiotensin II levels are going to be increased. Many clinical observations in COVID-19 have shown the high incidence of acute kidney injury that may be due to excessive levels of angiotensin II. The investigators hypothesize that administration of angiotensin (1-7) replaces levels of ACE-2 in COVID-19 and thereby ameliorates deterioration of multi-organ failure and specifically acute kidney injury.

ELIGIBILITY:
Inclusion Criteria:

* Severe COVID-19: Adult patients admitted to the hospital through the Emergency Department (ED) requiring oxygen therapy (any level) to maintain oxygen saturation (SaO2) > 90%
* COVID positive by polymerase chain reaction (PCR) on hospital admission
* Hospitalized patients aged 18 years or greater

Exclusion Criteria:

* Pre-existing chronic kidney disease
* New use of or change in dose of ACE-inhibitors or angiotensin receptor blocker (ARB) within the last 6 months
* Acute kidney injury at the time of enrollment defined as either increase pf serum creatinine by more than 50% or 0.3 mg/dL above baseline or estimated creatinine clearance (by MDRD) of less than 60 ml/min (if no baseline serum creatinine available)
* Pregnant and breastfeeding women
* Contraindicated medications: new use or change of medications from start of trial (start of an ACE inhibitor or ARB within 6 months of trial).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanine D'Armiento, MD, PhD, Principal Investigator — Associate Professor of Medicine in Anesthesiology
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Wagener G, Goldklang MP, Gerber A, Elisman K, Eiseman KA, Fonseca LD, D'Armiento JM. A randomized, placebo-controlled, double-blinded pilot study of angiotensin 1-7 (TXA-127) for the treatment of severe COVID-19. Crit Care. 2022 Jul 28;26(1):229. doi: 10.1186/s13054-022-04096-9. No abstract available. PMID 35902867

RESULTS

PARTICIPANT FLOW:
Groups:
- TXA127: Participants received one 3-hour dosage (0.5 mg/kg per day), intravenously, for 10 days consecutively (or until discharge if less than 10 days).
  TXA127: 0.5 mg/kg per day
- Placebo: Participants received one 3-hour dosage (0.5 mg/kg per day), intravenously, for 10 days consecutively (or until discharge if less than 10 days).
  Placebo: 0.5 mg/kg per day
Period: Overall Study
Arm/Group | TXA127 | Placebo
Started | 11 | 11
Completed | 6 | 9
Not Completed | 5 | 2
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Physician Decision | 2 | 1

BASELINE CHARACTERISTICS:
Population: We included in our analysis participants whom completed minimum of 1 day of drug/placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | TXA127 | Placebo | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Continuous [Mean (Full Range); unit: years] | 55 [41 to 79] | 55 [28 to 83] | 55 [28 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 9 | 4 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 7 | 15
  Not Hispanic or Latino | 3 | 1 | 4
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 9 | 20
Oxygen at randomization [Count of Participants; unit: Participants]
  Room air | 0 | 0 | 0
  Nasal cannula | 7 | 8 | 15
  High flow nasal cannula | 3 | 1 | 4
  Non-invasive ventilation/BiPAP | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change of Serum Creatinine
Description: Calculated from baseline (at enrollment) to end of study
Time Frame: Day 1 and Day 10
Population: Only subjects who received at least 1 complete dose of drug/placebo were included in the data analysis - which is not the same as those who "completed" the study as seen under Participant Flow. This included 11 out of 11 in the TXA127 group and 9 out of 11 in the Placebo group.
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | TXA127 | Placebo
Number analyzed (Participants) | 11 | 9
mg/dL | 0.92 [0.56 to 1.26] | 0.70 [0.45 to 1.11]

2. Primary Outcome: Number of Participants Requiring Intubation
Time Frame: From Day 1 to Day 10
Population: Only subjects who received at least 1 complete dose of drug/placebo were included in the data analysis. This included 11 out of 11 in the TXA127 group and 9 out of 11 in the Placebo group.
Measure: Count of Participants; unit: Participants
Arm/Group | TXA127 | Placebo
Number analyzed (Participants) | 11 | 9
Participants | 3 | 2

3. Secondary Outcome: Number of Participants Requiring Dialysis
Time Frame: Up to Day 10
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | TXA127 | Placebo
Number analyzed (Participants) | 11 | 9
Participants | 0 | 0

4. Secondary Outcome: Number of Participants Requiring a Vasopressors
Time Frame: Up to Day 10
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | TXA127 | Placebo
Number analyzed (Participants) | 11 | 9
Participants | 3 | 1

5. Secondary Outcome: Percent Change in Supplemental Oxygen Requirements
Time Frame: Day 1 and Day 10
Population: as for outcome 2
Measure: Mean (Full Range); unit: percent change of oxygen
Arm/Group | TXA127 | Placebo
Number analyzed (Participants) | 11 | 9
percent change of oxygen | 0.71 [-5.0 to 5.38] | 0.91 [-5.05 to 5.68]

6. Secondary Outcome: Days of Hospital Stay and Drug Administration
Time Frame: Day 1 to Day 10
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | TXA127 | Placebo
Number analyzed (Participants) | 11 | 9
days
  Length of Hospital Stay | 11 [6 to 21] | 7 [6 to 8]
  Days of Drug/placebo administration | 4 [2.5 to 8.5] | 5 [4 to 6]

7. Secondary Outcome: Cytokine Levels on the Day of Drug/TXA Administration
Time Frame: Day 1
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | TXA127 | Placebo
Number analyzed (Participants) | 10 | 9
pg/ml
  Interferon-γ | 1.44 [0.64 to 2.24] | 1.0 [0.59 to 1.32]
  IL-1β | 20.7 [11.7 to 41.9] | 30.6 [10.9 to 75.3]
  IL-1Ra | 15.9 [8.73 to 17.21] | 7.6 [4.48 to 19.19]
  IL-2 | 0.52 [0.19 to 1.17] | 0.37 [0.16 to 0.68]
  IL-4 | 0.41 [0.21 to 0.78] | 0.21 [0.05 to 1.79]
  IL-5 | 1.72 [1.02 to 8.20] | 1.21 [0.90 to 1.69]
  IL-6 | 9.63 [5.58 to 51.79] | 3.35 [2.79 to 9.53]
  IL-8 | 24.4 [15.9 to 61.1] | 16.2 [10.3 to 23.34]
  TNF-α | 68.4 [30.9 to 95.9] | 45.9 [37.16 to 58.7]
  IL-10 | 12.3 [5.4 to 29.6] | 10.8 [1.35 to 25.6]
  IL-12p40 | 32.4 [24.5 to 64.2] | 28.9 [18.1 to 45.4]
  IL-12p70 | 1.74 [0.83 to 2.74] | 0.63 [0.30 to 1.38]
  IL-13 | 9.9 [8.11 to 43.5] | 8.5 [6.49 to 14.2]
  MCP-1 | 345 [248 to 479] | 283 [219 to 351]

8. Secondary Outcome: Cytokine Levels on the Day 5 of Drug/TXA Administration
Time Frame: Day 5
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | TXA127 | Placebo
Number analyzed (Participants) | 5 | 4
pg/ml
  Interferon-γ | 0.88 [0.59 to 1.63] | 0.78 [0.58 to 1.06]
  IL-1β | 14.4 [6.1 to 27.0] | 50.6 [29.7 to 71.6]
  IL-1Ra | 17.77 [7.92 to 28.43] | 7.38 [4.18 to 16.78]
  IL-2 | 0.20 [0.12 to 0.48] | 0.91 [0.83 to 4.37]
  IL-4 | 0.09 [0.05 to 0.30] | 0.74 [0.44 to 1.04]
  IL-5 | 3.36 [2.34 to 11.74] | 0.99 [0.77 to 2.99]
  IL-6 | 12.88 [5.03 to 33.21] | 1.34 [0.78 to 6.89]
  IL-8 | 24.5 [14.1 to 29.3] | 14.3 [6.5 to 56.82]
  TNF-α | 31.1 [27.3 to 61.8] | 42.1 [36.2 to 60.4]
  IL-10 | 2.46 [2.03 to 2.75] | 4.19 [1.65 to 6.79]
  IL-12p40 | 45.40 [31.7 to 55.9] | 29.8 [22.1 to 38.9]
  IL-12p70 | 1.28 [0.42 to 1.64] | 1.21 [0.89 to 1.58]
  IL-13 | 10.71 [8.11 to 25.01] | 11.4 [11.1 to 13.9]
  MCP-1 | 218 [191 to 317] | 237 [179 to 264]

9. Secondary Outcome: Mortality
Time Frame: Day 1 to Day 10
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | TXA127 | Placebo
Number analyzed (Participants) | 11 | 9
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from Day 1 to Day 10 of study drug/placebo administration (or as long as hospitalized if less than 10 days) and at Day 28 and Day 60 (post hospital discharge) during a follow-up phone call.
Description: Only subjects who received at least 1 complete dose of drug/placebo were included in the data analysis - which is not the same as those who "completed" the study as seen under Participant Flow. This included 11 out of 11 in the TXA127 group and 9 out of 11 in the Placebo group.
Arm/Group | TXA127 | Placebo
All-Cause Mortality (participants affected / at risk) | 2/11 | 1/9
Serious Adverse Events (participants affected / at risk) | 3/11 | 2/9
Other Adverse Events (participants affected / at risk) | 7/11 | 5/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TXA127 (N=11) | Placebo (N=9)
Intubation (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TXA127 (N=11) | Placebo (N=9)
Right abdominal side pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diaphoresis (General disorders) | 0 (0) | 1 (1)
Refractory Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Refractory Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 2 (2) | 0 (0)
Vertigo (General disorders) | 0 (0) | 1 (1)
Hematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) — Blood in stool
Nausea (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Dyshidrotic Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Itchy hands and feet
Fever (General disorders) | 1 (1) | 0 (0)
Tussis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Angina Pectoris (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Chest Tightness
Cloudiness of Consciousness (General disorders) | 1 (1) | 0 (0) — Brain fog
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Transient Paresthesia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Numbness in left leg

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-25): https://cdn.clinicaltrials.gov/large-docs/23/NCT04401423/Prot_SAP_000.pdf